CLINICAL TRIAL: NCT03318731
Title: Evaluation of the Efficacy and Safety of Fenugreek Extract on Markers of Muscle Damage and Inflammation on Healthy Non-resistance Trained Participants
Brief Title: Efficacy and Safety of Fenugreek Extract on Markers of Muscle Damage and Inflammation in Untrained Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mary Hardin-Baylor (Other)
Collaborators: Indus Biotech Ltd. Pvt. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FNG-1
Record Dates: First submitted 2017-10-02; First posted 2017-10-24 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Muscle Damage; Inflammation
Keywords: fenugreek extract; non-resistance trained
MeSH Terms: conditions — Inflammation | interventions — Sugars; fenugreek seed meal

STUDY DESIGN:
Intervention Model Description: Three groups: placebo, 300mg dose (low) and 500mg dose (high)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sugar Pill (Placebo Comparator): Maltodextrin (matches the weight of the active treatment). Taken 1-hour prior to workout on training days and each day of overreaching week. On rest days, will consume in the morning with breakfast.
  Interventions: Other: Sugar Pill
- Fenugreek Extract, Low Dose (Experimental): 300mg Taken 1-hour prior to workout on training days and each day of overreaching week. On rest days, will consume in the morning with breakfast.
  Interventions: Dietary Supplement: Fenugreek Extract, Low Dose
- Fenugreek Extract, High Dose (Experimental): 500mg Taken 1-hour prior to workout on training days and each day of overreaching week. On rest days, will consume in the morning with breakfast.
  Interventions: Dietary Supplement: Fenugreek Extract, High Dose

INTERVENTIONS:
Other: Sugar Pill — Taken orally in capsule form
  Arms: Sugar Pill
Dietary Supplement: Fenugreek Extract, Low Dose — Taken orally in capsule form
  Arms: Fenugreek Extract, Low Dose
Dietary Supplement: Fenugreek Extract, High Dose — Taken orally in capsule form
  Arms: Fenugreek Extract, High Dose

SUMMARY:
This is a randomized, repeated measures and double blind study which measures the effect of fenugreek extract on markers of muscle damage and inflammation in non-resistance trained males. Participants will complete baseline testing and then be randomized into groups. Participants will complete a 2 week, split-body resistance training program. They will then return for testing in which they will complete an overreaching protocol for 5 consecutive days. Measurements will be recorded 24 hrs after the fifth day. Participants will resume the training program for one additional week and return for final measurements.

DETAILED DESCRIPTION:
Subjects expressing interest in doing the study will be interviewed in the UMHB Human Performance Lab (HPL) to determine whether they qualify to participate in the study. Upon qualification, participants will be scheduled a familiarization session in which they will be taught how to perform a proper bench press, back squat, deadlift and squat thruster. They will then schedule their first testing session which will include: a body composition analysis via an InBody 770, thigh circumference measurements, joint mobility measurements, a blood draw, strength testing (1RM), and muscular endurance testing (70% 1RM max reps). Participants will then be placed in groups based on fat free mass and assigned their workout program (3days/week) with training loads based on their 1RM values (bench press, back squat, deadlift and squat thruster).

Supplementation protocol: Participants will be randomly assigned into one of three groups and instructed to ingest capsules of either a placebo, or IND03 (fenugreek extract) containing 300mg, or 500mg. They will supplement 1 hour prior to their workout each exercise day as well as during the overreaching week. On "off/rest" days, participants will consume capsules in the morning with breakfast.

After two weeks of training, participants will return to the HPL for follow-up strength testing (1RM), and muscular endurance testing (70% 1RM max reps), then instructed to rest for 48 hours and return to the lab to begin their overreaching protocol. During each of the 5 days, participants undergo the following measurements prior to the exercise protocol: thigh circumference, joint mobility, and questionnaires (WOMAC & VAS). On Day 1 participants will also perform an InBody and blood draw. A blood draw will also be performed on Day 3. They will then consume a standardized snack and begin the overreaching protocol of 8 sets of 10 repetitions for the following 4 exercises: bench press, back squat, deadlift and squat thruster. There will be a 1 minute rest period in between each set and a 2 minute rest in between each exercise. Participants will then fill out a Rate of Perceived Exertion (RPE) immediately after the protocol. Again, they will perform this for 5 consecutive days.

Twenty-four hours after the last overreaching day, participants will return for thigh circumference, joint mobility, questionnaires (WOMAC & VAS), a blood draw, strength testing (1RM), and muscular endurance testing (70% 1RM max reps). They will then be instructed to continue the resistance training program for 1 week. After that period they will return for final measurements of thigh circumference, joint mobility, questionnaires (WOMAC & VAS), a blood draw, strength testing (1RM), and muscular endurance testing (70% 1RM max reps).

Throughout the duration of the study, participants will record their dietary intake via MyFitnessPal.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be males between the age of 18-45;
* Subjects will have not been participating in a structured resistance training program in the past 6 months;
* Subjects will be provided written and dated informed consent to participate in the study;
* Subjects will be willing and able to comply with the protocol;
* Subjects will be apparently healthy and free from disease, as determined by a health history questionnaire;
* Subjects will agree to abstain from exercise 48 hours prior to each testing visit;
* Subjects will agree to fast for 10 hours prior to each testing visit;
* Subjects will be agree to refrain from tobacco use, alcohol and/or caffeine consumption and/or smoking 12 hours prior to each testing visit;
* Subjects will agree to refrain from taking any supplement that may interfere with study supplementation for the remainder of the study.

Exclusion Criteria:

* Subject has taken ergogenic levels of nutritional supplements that may affect muscle mass (e.g., creatine, HMB) or anabolic/catabolic hormone levels (e.g., androstenedione, DHEA, etc.) within 3 months prior to the start of the study;
* Subject is unable to complete blood draws needed at each testing session;
* Subject reports any unusual adverse events associated with this study that in consultation with the supervising physician recommends removal from the study;
* Subject does not complete 90% of resistance training program assigned;
* Subject is unable to complete overreaching protocol during overreaching week;

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Effect of Fenugreek Extract on Interleukin-1 | within 26 days
  The primary purpose of this investigation is to determine the effectiveness of fenugreek extract on blunting an exercise-induced state of inflammation during a period of high volume and overreaching resistance exercise in young, non-resistance trained males. This will be accomplished by observing blood markers prior to, during and post exercise testing.
Effect of Fenugreek Extract on Creatine Kinase | within 26 days
  The primary purpose of this investigation is to determine if supplementation of fenugreek extract will have a protective effect on muscle damage in response to resistance exercise. This will be accomplished by observing blood markers prior to, during and post exercise testing.
Effect of Fenugreek Extract on Interleukin-6 | within 26 days
  The primary purpose of this investigation is to determine the effectiveness of fenugreek extract on blunting an exercise-induced state of inflammation during a period of high volume and overreaching resistance exercise in young, non-resistance trained males. This will be accomplished by observing blood markers prior to, during and post exercise testing.
Effect of Fenugreek Extract on Tumor Necrosis Factor Alpha (TNF-α) | within 26 days
  The primary purpose of this investigation is to determine the effectiveness of fenugreek extract on blunting an exercise-induced state of inflammation during a period of high volume and overreaching resistance exercise in young, non-resistance trained males. This will be accomplished by observing blood markers prior to, during and post exercise testing.
Effect of Fenugreek Extract on C-reactive protein | within 26 days
  The primary purpose of this investigation is to determine the effectiveness of fenugreek extract on blunting an exercise-induced state of inflammation during a period of high volume and overreaching resistance exercise in young, non-resistance trained males. This will be accomplished by observing blood markers prior to, during and post exercise testing.
Effect of Fenugreek Extract on 3-methylhistidine | within 26 days
  The primary purpose of this investigation is to determine if supplementation of fenugreek extract will have a protective effect on muscle damage in response to resistance exercise. This will be accomplished by observing blood markers prior to, during and post exercise testing.
Effect of Fenugreek Extract on Lactate Dehydrogenase | within 26 days
  The primary purpose of this investigation is to determine if supplementation of fenugreek extract will have a protective effect on muscle damage in response to resistance exercise. This will be accomplished by observing blood markers prior to, during and post exercise testing.

SECONDARY OUTCOMES:
Effect of Fenugreek Extract on Glucose mg/dL | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Urea Nitrogen (BUN) mg/Dl | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Creatinine mg/Dl | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on eGFR Non-Afr. American mL/min/1.73m2 | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on eGFR African American mL/min/1.73m2 | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on BUN/Creatinine Ratio calculated | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Sodium mmol/L | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Potassium mmol/L | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Chloride mmol/L | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Carbon Dioxide mmol/L | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Calcium mg/Dl | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Protein, Total g/Dl | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Albumin g/dL | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Globulin g/Dl | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Albumin/Globulin Ratio calculated | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Bilirubin, Total mg/Dl | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Alkaline Phosphatase U/L | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Aspartate Aminotransferase U/L | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Alanine Aminotransferase U/L | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a comprehensive metabolic panel prior to and after the supplementation period.
Effect of Fenugreek Extract on White Blood Cell Count thousand/uL | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Red Blood Cell Count million/uL | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Hemoglobin g/dL | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Hematocrit % | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on MCV fL | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on MCH pg | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on MCHC g/dL | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on RDW % | within 26 days
  v
Effect of Fenugreek Extract on Platelet Count thousand/uL | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on MPV fL | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Absolute Neutrophils cells/uL | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Absolute Lymphocytes cells/uL | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Absolute Monocytes cells/uL | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Absolute Eosinophils cells/uL | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Absolute Basophils cells/uL | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Neutrophils % | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Lymphocytes % | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Monocytes % | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Eosinophils % | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.
Effect of Fenugreek Extract on Basophils % | within 26 days
  The secondary purpose is to assess safety of ingestion of the supplement with analysis of a complete blood count panel prior to and after the supplementation period.

CONTACTS AND LOCATIONS:
Overall Officials: Lemuel W Taylor IV, PhD, Principal Investigator — UMHB Human Performance Lab
Locations (1):
- UMHB Human Performance Lab, Belton, Texas, United States

IPD SHARING:
Plan to Share IPD: No